CLINICAL TRIAL: NCT00728832
Title: A Phase 1 Study to Evaluate the Effects of Lidocaine/Epinephrine Test Dose Administration on the Pharmacokinetic Profile of a Single Dose of Thoracic Extended-Release Epidural Morphine in Patients Undergoing Major Upper Abdominal Surgery
Brief Title: A Pharmacokinetic (PK) Study of Extended-Release Epidural Morphine in Upper Abdominal Surgery
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: EKR Therapeutics, Inc (Industry)
Collaborators: Pacira Pharmaceuticals, Inc (Industry)
Responsible Party: Eugene R. Viscusi, MD, Thomas Jefferson University
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: SKY0401-016
Record Dates: First submitted 2008-08-01; First posted 2008-08-06 (Estimated); Last update posted 2008-08-14 (Estimated); Status verified 2008-08

CONDITIONS: Postoperative Pain
Keywords: extended release epidural morphine; morphine; thoracic epidural; pharmacokinetics; pharmacodynamics; postoperative pain; upper abdominal surgery
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- 1 (Active Comparator): No test dose + DepoDur + flush with 1 mL normal saline
  Interventions: Drug: DepoDur (extended-release epidural morphine)
- 2 (Experimental): Test dose + flush with 1 mL normal saline + 3-minute wait + DepoDur + flush with 1 mL normal saline
  Interventions: Drug: DepoDur (extended-release epidural morphine)
- 3 (Experimental): Test dose + flush with 1 mL normal saline + 10-minute wait + DepoDur + flush with 1 mL normal saline
  Interventions: Drug: DepoDur (extended-release epidural morphine)
- 4 (Experimental): Test dose + flush with 1 mL normal saline + 15-minute wait + DepoDur + flush with 1 mL normal saline
  Interventions: Drug: DepoDur (extended-release epidural morphine)
- 5 (Experimental): Test dose + No flush + 3-minute wait + DepoDur + flush with 1 mL normal saline
  Interventions: Drug: DepoDur (extended-release epidural morphine)

INTERVENTIONS:
Drug: DepoDur (extended-release epidural morphine) — DepoDur with on demand boluses of IV fentanyl PCA

SUMMARY:
The primary purpose of this study is to evaluate the effects of lidocaine/epinephrine test dose administration on the PK profile of a single epidural dose of DepoDur (extended-release epidural morphine) in patients undergoing major upper abdominal surgery. A secondary objective was to evaluate the safety and efficacy profile.

ELIGIBILITY:
Inclusion Criteria:

* Males and females ≥ 18 years of age at Screening
* Negative pregnancy test in females of childbearing potential
* Scheduled for major upper abdominal surgery via an upper midline incision under general anesthesia
* American Society of Anesthesiology (ASA) Physical Class 1, 2, or 3
* Willing and able to use a PCA pump
* Willing to receive only IV fentanyl for 72 hours post-dose to control post-operative pain
* Capable of providing written informed consent and responses to pain assessment scales and neurological assessment questionnaires

Exclusion Criteria:

* Morbid obesity, defined as a body mass index (BMI) ≥ 40
* Scheduled to undergo surgery under regional anesthesia
* Usage of analgesic medications containing morphine or codeine within three days prior to study drug administration
* Chronic opioid medication usage (defined as daily opioids for more than 7 days prior to enrollment)
* Suspected or documented history of sleep apnea, narcolepsy, or excessive daytime sleepiness
* Female who was pregnant or lactating
* History of hypersensitivity or idiosyncratic reaction to opioid medications, local anesthetics, or epinephrine
* Any contraindication for the epidural administration of study drug (e.g., coagulopathy, local infection)
* Administration of an investigational drug within 30 days prior to Screening
* Suspected or documented history of substance abuse and/or alcoholism
* Any contraindication to frequent blood PK sampling (such as significant anemia) or other barrier to obtaining timely PK samples

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2002-05; Primary Completion 2003-02 (Actual)

PRIMARY OUTCOMES:
Evaluate the serum pharmacokinetic profile of a single 15-mg dose of DepoDur administered at the lower thoracic epidural space with or without a prior lidocaine-epinephrine test dose

SECONDARY OUTCOMES:
efficacy and safety profiles

CONTACTS AND LOCATIONS:
Overall Officials: Eugene R Viscusi, MD, Principal Investigator — Thomas Jefferson University

REFERENCES:
- [Derived] Viscusi ER, Manvelian GZ. A randomized study of the serum pharmacokinetics of lower thoracic extended-release epidural morphine (DepoDur) after lidocaine-epinephrine test dose administration in patients undergoing upper abdominal surgery. Int J Clin Pharmacol Ther. 2009 Nov;47(11):659-70. doi: 10.5414/cpp47659. PMID 19840530